CLINICAL TRIAL: NCT04930107
Title: Prospective Studies of Vaginal Yeast and Microbiome Related to Vulvovaginal Candidiasis in Canadian Females
Brief Title: Vulvovaginal Candidiasis in Canadian Females
Acronym: THRIVE-yeast
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Medical Service Foundation (Other); Research Manitoba (Other)
Responsible Party: Principal Investigator, Aleeza Gerstein, Assistant Professor, University of Manitoba
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B2021:026
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Candidiasis, Vulvovaginal
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Fluconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Recurrent Infection Cohort - symptomatic (Active Comparator): Participants with a history of recurrent vulvovaginal candidiasis infections who have an active symptomatic infection when they come to clinic
  Interventions: Drug: Fluconazole 150 mg; Drug: Boric Acid Supp,Vag
- Asymptomatic Cohort (No Intervention): Participants with no history of vulvovaginal candidiasis
- Recurrent Infection Cohort - asymptomatic (No Intervention): Participants with a history of recurrent vulvovaginal candidiasis infections who do not have an active symptomatic infection when they come to clinic

INTERVENTIONS:
Drug: Fluconazole 150 mg — Treatment will be offered to participants if clinical exam and clinical samples are consistent with vulvovaginal candidiasis (VVC). Females presenting with a suspected first-time yeast infection will be treated with fluconazole 150 mg orally.
  Arms: Recurrent Infection Cohort - symptomatic
Drug: Boric Acid Supp,Vag — Treatment will be offered to participants if clinical exam and clinical samples are consistent with vulvovaginal candidiasis (VVC). Women that have had a prior documented VVC infection that has recurred on fluconazole will be treated with boric acid, 600 mg intravaginally at bedtime for 7 days.
  Arms: Recurrent Infection Cohort - symptomatic

SUMMARY:
Vulvovaginal candidiasis (VVC; colloquially referred to as a 'yeast infection') is a prevalent mucosal infection caused by Candida spp. that affects ~75% of women at least once in their life. VVC usually responds well to treatment, yet a small but significant fraction of women experience recurrent yeast infections even with weekly treatment. A further complication in understanding the causes of recurrent infections is that approximately one in five females have vaginal yeast present without any symptoms at any given point. The link between fungi, other microbes in the vagina ("microbiome"), and the human immune system remain poorly understood in the switch from having yeast present in the vagina without any symptoms and symptomatic yeast infections. Fungi also compose a normal component of the microbiome at other sites in the body (e.g., oral, skin, gastrointestinal tract, rectum) where they may serve as a source of re-infection following treatment.

In addition to the commonly prescribed 'first choice' antifungal drug fluconazole, a second-line treatment, boric acid, has shown promise in the literature and has been used locally with success at increasing the time between recurrent infections. A drawback of this therapy, however, is cost, as it is a compounded medication, and patients have to pay out of pocket. The purpose of this study is to understand how the yeast and bacterial microbial communities differ for females with recurrent infections from females with their first yeast infection and females with vaginal yeast present without any symptoms, and to track yeast diversity following treatment with either boric acid or fluconazole. The investigators hypothesize that they will identify multiple subpopulations of yeast at multiple anatomical body sites in females with VVC and recurrent VVC. They anticipate finding evidence for recurrent infection from secondary sites by linking genomic diversity of vaginal yeast strains during symptomatic infection to strains from other body sites. They hypothesize that yeast isolated from females with recurrent infections will exhibit different drug response phenotypes than yeast from females with asymptomatic vaginal yeast. They hypothesize that the vaginal microbiome of post-treatment patients treated with boric acid will differ from that of fluconazole. Combined, they hypothesize that post-treatment response will differ between the drugs, indicating that treatment specifics influence the vaginal environment.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between ages of 18 and 50 years.

Exclusion Criteria:

* Currently pregnant
* Trying to get pregnant
* Have had a hysterectomy
* BV infection

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Fungal Diversity | One month
  Use culture-based methods, flow cytometry, and genome sequencing to:
  * Test how genotypic diversity, genetic relatedness, and drug resistance and tolerance changes in the fungal population from the assumed first-time infection cohort and recurrent infection cohort participants before and after treatment with either fluconazole or boric acid.
  * How the vaginal fungal population diversity differs between symptomatic and asymptomatic participants.
  * Test how the vaginal fungal isolates in participants with VVC are related to rectal, oral, and skin fungal isolates.

SECONDARY OUTCOMES:
Bacterial Diversity | One month
  Using 16S-rRNA sequencing and meta-proteomic to characterize the bacterial diversity changes pre-and post- drug treatment for VVC.
Host Functional Changes | One month
  Host proteome of the vaginal samples will be assessed using proteomics to determine any underlying inflammatory or barrier pathways that associate with treatment of VVC.

CONTACTS AND LOCATIONS:
Overall Officials: Aleeza Gerstein, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Health Science Centre (HSC), Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified proteomics and microbiome data collected will be placed into a freely available data repository after peer review of publications via Genbank. The proteomic expression data shall be made available by depositing the raw, untransformed and normalized counts on our servers. Whole genome sequencing data will be made available on the National Center for Biotechnology Information (NCBI) short reads archive. Any other functional data shall be made available with the journal publications in the text, or as supplementary material at the publisher's online website, or in data repositories (e.g., Dryad, https://datadryad.org).
Supporting Information: Analytic Code
Time Frame: Following publication in peer-reviewed journal articles, data available indefinitely.
Access Criteria: Following publication, external collaborators wishing to make use of THRIVE-yeast data must first contact the PI and submit a written proposal to request access to de-identified data. The PI will consult with University of Manitoba Office of Research Services to create a Data Sharing Transfer Agreement.